CLINICAL TRIAL: NCT05465460
Title: Effect of Banana Blossom on Breast Milk Volume in Mothers of Preterm Newborns, a Randomized, Double Blinded, Placebo-controlled Trial
Brief Title: Effect of Banana Blossom on Breast Milk Volume in Mothers of Preterm Newborns
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Vorapong Phupong, Prof. Vorapong Phupong, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 667/2022
Record Dates: First submitted 2022-07-07; First posted 2022-07-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Preterm Birth; Postpartum Women
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Banana blossom (Active Comparator): Participants received banana blossom 225 mg tablet orally four time per day for 14 days.
  Interventions: Drug: Banana Blossom
- Placebo (Placebo Comparator): Participants received placebo tablet orally four time per day for 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Banana Blossom — Banana Blossom 225 mg tablet orally four times per day for 14 days
  Arms: Banana blossom
Drug: Placebo — Placebo tablet orally four times per day for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effect of banana blossom in increasing breast milk volume

ELIGIBILITY:
Inclusion Criteria:

* Postpartum women of preterm newborns

Exclusion Criteria:

* Postpartum women with contraindication for breast feeding such as HIV, herpes zoster at breast, infected wound at breast.
* Postpartum women with preeclampsia, diabetes mellitus, postpartum hemorrhage.
* Postpartum women with allergy to banana blossom.
* Postpartum women with previous breast surgery or nipple surgery.
* Postpartum women who smoking.
* Preterm newborns with unstable conditions.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Breast milk volume per day at day 14 | at day 14
  Breast milk volume measurement in milliliters
Breast milk volume per day at day 3 | at day 3
  Breast milk volume measurement in milliliters
Breast milk volume per day at day 7 | at day 7
  Breast milk volume measurement in milliliters

SECONDARY OUTCOMES:
percentage of good satisfaction | at 14 days
  satisfaction evaluated by 5 Likert scales
percentage of side effects during intervention | day 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14
  percentage of participants with side effects such as headache, nausea/vomiting assessing by asking
percentage of drug compliance | at 14 days
  percentage of complete drug use assessing by remained drug counting
factors associated with increasing breast milk volume | at 14 days
  factors associated with increasing breast milk volume assessing by univariate and multivariate analysis

CONTACTS AND LOCATIONS:
Overall Officials: Vorapong Phupong, M.D., Study Director — Chulalongkorn University, Faculty of Medicine, Department of Obstetrics and Gynecology
Locations (1):
- Vorapong Phupong, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hill PD, Aldag JC, Chatterton RT, Zinaman M. Comparison of milk output between mothers of preterm and term infants: the first 6 weeks after birth. J Hum Lact. 2005 Feb;21(1):22-30. doi: 10.1177/0890334404272407. PMID 15681632
- [Background] Yu X, Li J, Lin X, Luan D. Association between Delayed Lactogenesis Ⅱ and Early Milk Volume among Mothers of Preterm Infants. Asian Nurs Res (Korean Soc Nurs Sci). 2019 May;13(2):93-98. doi: 10.1016/j.anr.2019.02.001. Epub 2019 Feb 16. PMID 30776448
- [Background] Ronnestad A, Abrahamsen TG, Medbo S, Reigstad H, Lossius K, Kaaresen PI, Egeland T, Engelund IE, Irgens LM, Markestad T. Late-onset septicemia in a Norwegian national cohort of extremely premature infants receiving very early full human milk feeding. Pediatrics. 2005 Mar;115(3):e269-76. doi: 10.1542/peds.2004-1833. Epub 2005 Feb 1. PMID 15687416
- [Background] Lai CT, Hale TW, Simmer K, Hartmann PE. Measuring milk synthesis in breastfeeding mothers. Breastfeed Med. 2010 Jun;5(3):103-7. doi: 10.1089/bfm.2009.0074. PMID 20433368
- [Background] Amornlerdpison D CV, Narkprasom K, Yimyam S. Bioactive Compounds and Antioxidant Properties of Banana Inflorescence in a Beverage for Maternal Breastfeeding. Applied Sciences. 2020; 11(1):343.
- [Background] Koduri PB, Rillema JA. Saponin effects of prolactin-like stimulation of ornithine decarboxylase activity in mouse mammary gland explants. Horm Metab Res. 1992 Dec;24(12):562-4. doi: 10.1055/s-2007-1003390. PMID 1478613
- [Background] Mathew NS, Negi PS. Traditional uses, phytochemistry and pharmacology of wild banana (Musa acuminata Colla): A review. J Ethnopharmacol. 2017 Jan 20;196:124-140. doi: 10.1016/j.jep.2016.12.009. Epub 2016 Dec 14. PMID 27988402
- [Background] Mahmood A, Omar MN, Ngah N. Galactagogue effects of Musa x paradisiaca flower extract on lactating rats. Asian Pac J Trop Med. 2012 Nov;5(11):882-6. doi: 10.1016/S1995-7645(12)60164-3. PMID 23146802
- [Background] Slusher T, Slusher IL, Biomdo M, Bode-Thomas F, Curtis BA, Meier P. Electric breast pump use increases maternal milk volume in African nurseries. J Trop Pediatr. 2007 Apr;53(2):125-30. doi: 10.1093/tropej/fml066. PMID 17409102
- [Background] Jones E, Dimmock PW, Spencer SA. A randomised controlled trial to compare methods of milk expression after preterm delivery. Arch Dis Child Fetal Neonatal Ed. 2001 Sep;85(2):F91-5. doi: 10.1136/fn.85.2.f91. PMID 11517200
- [Background] Geddes D, Hartmann P, Jones E. Preterm birth: Strategies for establishing adequate milk production and successful lactation. Semin Fetal Neonatal Med. 2013 Jun;18(3):155-159. doi: 10.1016/j.siny.2013.04.001. Epub 2013 Apr 26. PMID 23623976
- [Result] Foong SC, Tan ML, Foong WC, Marasco LA, Ho JJ, Ong JH. Oral galactagogues (natural therapies or drugs) for increasing breast milk production in mothers of non-hospitalised term infants. Cochrane Database Syst Rev. 2020 May 18;5(5):CD011505. doi: 10.1002/14651858.CD011505.pub2. PMID 32421208
- [Result] Nordin ZM BI, Omar MN, Mahmood A. Effect of consuming lactogenic biscuits formulated with banana (Musa x paradisiaca) flower flour on expressed breast milk (EBM) among lactating working women. Food Research 2019;4(2):294-300.
- [Result] Khorana M, Wongsin P, Torbunsupachai R, Kanjanapattanakul W. Effect of Domperidone on Breast Milk Production in Mothers of Sick Neonates: A Randomized, Double-Blinded, Placebo-Controlled Trial. Breastfeed Med. 2021 Mar;16(3):245-250. doi: 10.1089/bfm.2020.0234. Epub 2020 Nov 17. PMID 33202169